CLINICAL TRIAL: NCT01749930
Title: A Randomized, Multicenter, Double-Masked, Parallel-Group Study Comparing the Safety and Efficacy of BOL-303259-X Ophthalmic Solution With Timolol Maleate Ophthalmic Solution 0.5% in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Comparing the Safety and Efficacy of BOL-303259-X Ophthalmic Solution With Timolol Maleate Ophthalmic Solution in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Acronym: LUNAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 770
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — BOL 303259-X; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOL-303259-X (Experimental): BOL-303259-X ophthalmic solution QD (PM) and vehicle QD (AM) administered for 3 months (Visit 6) into the study eye(s).
  Interventions: Drug: BOL-303259-X
- Timolol (Active Comparator): Timolol maleate ophthalmic solution, 0.5%, administered BID for 3 months (Visit 6) into study eye(s).
  Interventions: Drug: Timolol; Drug: BOL-303259-X

INTERVENTIONS:
Drug: BOL-303259-X — BOL-303259-X will be administered QD in the evening and its vehicle administered QD in the morning
  Arms: BOL-303259-X
Drug: Timolol — Timolol will be administered BID once in the morning and once in the evening.
  Arms: Timolol
Drug: BOL-303259-X — All participants will receive a topical ocular BOL-303259-X QD in the evening from 3 months (Visit 6) through 6 months (Visit7).

SUMMARY:
In participants with a diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT), the primary objective is to demonstrate that the mean IOP reduction after 3 months of treatment with BOL-303259-X once daily (QD) is non-inferior to timolol maleate 0.5% twice daily (BID). The secondary objective is to demonstrate the superiority of BOL-303259-X QD to timolol maleate 0.5% BID. This assessment will be performed if the non-inferiority of BOL-303259-X QD to timolol maleate 0.5% BID is determined. An open label safety phase will be conducted at the end of Visit 6 (3 months) where all participants will receive BOL-303259-X QD for an additional 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of OAG (including pigmentary or pseudoexfoliative) or OHT in 1 or both eyes.
* Participants must meet the following IOP requirements at Visit 3
* mean/median IOP ≥ 24 mmHg at a minimum of 2 time points in the same eye
* IOP ≤ 36 mmHg at all 3 measurement time points in both eyes.
* Participants with a best-corrected visual acuity (BCVA), using the Early Treatment of Diabetic Retinopathy Study (ETDRS) protocol, of +0.7 logMAR units (Snellen equivalent of approximately 20/100) or better in either eye.

Exclusion Criteria:

* Participants with known hypersensitivity or contraindications to latanoprost, NO treatment, timolol maleate, other beta-adrenergic receptor antagonists or any of the ingredients in the study drugs.
* Participants with a central corneal thickness greater than 600 μm in either eye.
* Participants with advanced glaucoma and participants with a cup/disc ratio greater than 0.8 or a history of split fixation, or a field loss threatening fixation in either eye.
* Participants who do not have an intact posterior capsule in either eye .
* Participants with aphakia in either eye.
* Participants with previous or active corneal disease in either eye.
* Participants with current or a history of severe dry eye in either eye.
* Participants with current or a history of optic disc hemorrhage in either eye.
* Participants with current or a history of central/branch retinal vein or artery occlusion in either eye.
* Participants with current or a history of macular edema in either eye.
* Participants with very narrow angles (3 quadrants with less than Grade 2 according to Shaffer's anterior chamber angle grading system) and participants with angle closure,congenital, and secondary glaucoma, and participants with history of angle closure in either eye.
* Participants with a diagnosis of a clinically significant or progressive retinal disease in either eye.
* Participants with any intraocular infection or inflammation in either eye within 3 months(90 days) prior to Visit 1 (Screening).
* Participants with a history of ocular laser surgery in either eye within the 3 months(90 days) prior to Visit 1 (Screening).
* Participants with a history of incisional ocular surgery or severe trauma in either eye within 3 months (90 days) prior to Visit 1 (Screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Vittitow, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Inc., Rochester, New York, United States

REFERENCES:
- [Result] Medeiros FA, Martin KR, Peace J, Scassellati Sforzolini B, Vittitow JL, Weinreb RN. Comparison of Latanoprostene Bunod 0.024% and Timolol Maleate 0.5% in Open-Angle Glaucoma or Ocular Hypertension: The LUNAR Study. Am J Ophthalmol. 2016 Aug;168:250-259. doi: 10.1016/j.ajo.2016.05.012. Epub 2016 May 20. PMID 27210275
- [Result] Weinreb RN, Liebmann JM, Martin KR, Kaufman PL, Vittitow JL. Latanoprostene Bunod 0.024% in Subjects With Open-angle Glaucoma or Ocular Hypertension: Pooled Phase 3 Study Findings. J Glaucoma. 2018 Jan;27(1):7-15. doi: 10.1097/IJG.0000000000000831. PMID 29194198

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BOL-303259-X | Timolol
Started | 283 (randomized population) | 137 (randomized population)
Completed | 253 (randomized population) | 125 (randomized population)
Not Completed | 30 | 12

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population. Of the 420 subjects randomized, 5 subjects did not receive any instillation of study medication. The safety population consisted of 415 subjects, whereas the ITT population consisted of 414 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | BOL-303259-X | Timolol | Total
Number analyzed (Participants) | 278 | 136 | 414
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (9.77) | 64.1 (9.71) | 64.7 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 79 | 241
  Male | 116 | 57 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 19 | 55
  Not Hispanic or Latino | 242 | 117 | 359
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 69 | 46 | 115
  White | 204 | 89 | 293
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean IOP
Description: Mean intraocular pressure (IOP) in the study eye measured at the specified time points: 8 AM, 12 PM, and 4 PM at Visit 4 (Week 2), Visit 5 (Week 6), and Visit 6 (Month 3).
Time Frame: 8 AM, 12 PM, and 4 PM at Visit 4 (Week 2), Visit 5 (Week 6), and Visit 6 (Month 3)
Population: Intent-to-treat population with LOCF
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Groups:
- BOL-303259-X: BOL-303259-X ophthalmic solution QD (PM) and vehicle QD (AM) administered for 3 months into the study eye.
- Timolol: Timolol maleate ophthalmic solution, 0.5%, administered BID for 3 months into study eye.
Arm/Group | BOL-303259-X | Timolol
Number analyzed (Participants) | 277 | 135
mm Hg
  8 am week 2: number analyzed (Participants) | 275 | 134
  8 am week 2 | 19.17 (3.748) | 19.61 (3.092)
  12 pm week 2: number analyzed (Participants) | 270 | 134
  12 pm week 2 | 18.46 (3.327) | 19.22 (3.241)
  4 pm week 2: number analyzed (Participants) | 270 | 134
  4 pm week 2 | 18.10 (3.135) | 18.79 (3.022)
  8 am week 6 | 18.67 (3.272) | 19.59 (3.324)
  12 pm week 6: number analyzed (Participants) | 271 | 135
  12 pm week 6 | 18.02 (3.073) | 18.86 (3.169)
  4 pm week 6: number analyzed (Participants) | 271 | 135
  4 pm week 6 | 17.87 (3.114) | 18.85 (3.415)
  8 am Month 3 | 18.68 (3.195) | 19.56 (3.318)
  12 pm Month 3: number analyzed (Participants) | 271 | 135
  12 pm Month 3 | 17.92 (3.119) | 19.21 (3.129)
  4 pm Month 3: number analyzed (Participants) | 271 | 135
  4 pm Month 3 | 17.72 (3.153) | 19.06 (3.002)
Statistical Analysis 1: Comparison: BOL-303259-X vs Timolol; Test type: Non-Inferiority — The 2 treatments were compared for each time point by visit. LS mean of each treatment group, the difference in the LS mean, and the 2-sided 95% CI for the difference were obtained. Noninferiority could be claimed if the upper limit of the CIs <1.5 mmHg at all time points of each visit and <1.00 mmHg for at least 5 out of the 9 time points. If noninferiority was determined, superiority at each time point could be claimed if the upper limit of the 95% CI<0 mmHg at all time points of each visit; p = 0.216, ANCOVA — The ANCOVA results for the comparison of LS means of mean IOP between treatment groups demonstrated noninferiority of BOL-303259-X to timolol. Superiority of BOL-303259-X to timolol was demonstrated at 8 of 9 time points (exception at 8 am Week 2)

2. Secondary Outcome: IOP ≤ 18 mm Hg
Description: Percentage of participants with IOP ≤ 18 mm Hg consistently at all 9 time points in the first 3 months
Time Frame: 8 AM, 12 PM, and 4 PM at Visit 4 (Week 2), Visit 5 (Week 6), and Visit 6 (Month 3)
Population: Intent-to treat population with LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | BOL-303259-X | Timolol
Number analyzed (Participants) | 277 | 135
Participants | 49 | 15
Statistical Analysis 1: Comparison: BOL-303259-X vs Timolol; Test type: Other; p = 0.084, Chi-squared

3. Secondary Outcome: IOP Reduction ≥ 25%
Description: Percentage of participants with IOP reduction ≥ 25% consistently at all 9 time points in the first 3 months
Time Frame: 8 AM, 12 PM, and 4 PM at Visit 4 (Week 2), Visit 5 (Week 6), and Visit 6 (Month 3)
Population: Intent-to-treat population with LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | BOL-303259-X | Timolol
Number analyzed (Participants) | 277 | 135
Participants | 86 | 25
Statistical Analysis 1: Comparison: BOL-303259-X vs Timolol; Test type: Other; p = 0.007, Chi-squared

4. Other Pre Specified Outcome: Number of Participants With Ocular and Systemic Adverse Events
Description: Following assessments through 3 months (Visit 6), all participants, irrespective of previous randomization, converted to a single open label safety arm receiving BOL-303259-X QD in the evening for an additional 3 months through Visit 7. Adverse events were recorded throughout the comparative efficacy phase and open label extension phase.
Time Frame: 6 months
Population: Safety population. Of the subjects randomized, 415 instilled at least one dose of study medication and were included in the safety population
Measure: Count of Participants; unit: Participants
Groups:
- BOL-303259-X: BOL-303259-X ophthalmic solution QD (PM) and vehicle QD (AM) administered for 3 months into the study eye during the efficacy phase
- Timolol: Timolol maleate ophthalmic solution, 0.5%, administered BID for 3 months into study eye during the efficacy phase
- BOL-303259-X Safety Extension Phase: Following completion of the efficacy phase, all subjects were converted to BOL-303259-X ophthalmic solution QD (PM) and vehicle QD (AM) for an additional 3 months during the open label safety extension phase
Arm/Group | BOL-303259-X | Timolol | BOL-303259-X Safety Extension Phase
Number analyzed (Participants) | 279 | 136 | 384
Participants
  >/= 1 nonocular AE | 36 | 18 | 23
  >/= 1 ocular (Study eye) AE | 66 | 18 | 53
Statistical Analysis 1: Comparison: BOL-303259-X vs Timolol; Test type: Other; No statistical analysis was performed on these proportions

ADVERSE EVENTS:
Time Frame: 6 months
Description: Safety Population (analyzed as treated). Of the subjects randomized, 415 instilled at least one dose of study medication and were included in the safety population.
  All subjects were converted to BOL-303259-X during the safety extension phase and AEs reported during that phase are presented below as a third arm.
Groups:
- BOL-303259-X Safety Extension Phase: Following completion of the efficacy phase, all subjects were converted to BL-303259-X ophthalmic solution QD (PM) and vehicle QD (AM) for an additional 3 months during the open label extension phase
Arm/Group | BOL-303259-X | Timolol | BOL-303259-X Safety Extension Phase
Serious Adverse Events (participants affected / at risk) | 4/279 | 0/136 | 2/384
Other Adverse Events (participants affected / at risk) | 50/279 | 12/136 | 32/384
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOL-303259-X (N=279) | Timolol (N=136) | BOL-303259-X Safety Extension Phase (N=384)
left shoulder subluxation of acromioclavicular joint (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scapular fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Uncontrolled hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelethiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Other convulsions (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in joint (shoulder) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subdural hermorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Closed dislocation of finger (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Closed fracture of distal end of ulna (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOL-303259-X (N=279) | Timolol (N=136) | BOL-303259-X Safety Extension Phase (N=384)
Conjunctival hyperemia (Eye disorders) | 25 (32) | 1 (1) | 18 (19)
Eye irritation (Eye disorders) | 20 (20) | 6 (7) | 8 (8)
Eye pain (Eye disorders) | 16 (16) | 5 (6) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No